CLINICAL TRIAL: NCT00964418
Title: A Trial Investigating the Pharmacodynamic and Pharmacokinetic Properties of NN1250 in Young and Geriatric Subjects With Type 1 Diabetes
Brief Title: A Trial Investigating the Effect of NN1250 in Young and Elderly Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-1994; 2008-008601-21 (EudraCT Number)
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg (Experimental)
  Interventions: Drug: insulin degludec
- IGlar (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — 0.4 U/kg body weight injected s.c. (subcutaneously) once daily for 6 days
  Arms: IDeg
Drug: insulin glargine — 0.4 U/kg body weight injected s.c. (subcutaneously) once daily for 6 days
  Arms: IGlar

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate the blood glucose lowering effect of NN1250 (insulin degludec) in young and elderly subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-35 years (both inclusive) (young group) or at least 65 years (geriatric group)
* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index 18.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve during one dosing interval at steady state (for NN1250) | 0-24 hours (derived on treatment day 6)

SECONDARY OUTCOMES:
Area under the NN1250 concentration-time curve during one dosing interval at steady state | 0-24 hours (derived on treatment day 6)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

REFERENCES:
- [Result] Korsatko S, Deller S, Mader JK, Glettler K, Koehler G, Treiber G, Urschitz M, Wolf M, Hastrup H, Sondergaard F, Haahr H, Pieber TR. Ultra-long pharmacokinetic properties of insulin degludec are comparable in elderly subjects and younger adults with type 1 diabetes mellitus. Drugs Aging. 2014 Jan;31(1):47-53. doi: 10.1007/s40266-013-0138-0. PMID 24263619
- [Result] Heise T, Korsatko S, Nosek L, Coester HV, Deller S, Roepstorff C, Segel S, Kapur R, Haahr H, Hompesch M. Steady state is reached within 2-3 days of once-daily administration of degludec, a basal insulin with an ultralong duration of action. J Diabetes. 2016 Jan;8(1):132-8. doi: 10.1111/1753-0407.12266. Epub 2015 Mar 24. PMID 25581159
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com